CLINICAL TRIAL: NCT00123214
Title: Pilot Study: A Dietary Intervention May Decrease the Negative Metabolic and Cognitive Consequences of Chronic Sleep Deprivation
Brief Title: A Change in Diet May Decrease the Negative Consequences of Chronic Sleep Deprivation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Vincent's Medical Center (Unknown)
Collaborators: Inflammation Research Foundation, Marblehead, MA. (Unknown); NeuroScience, Inc., Osceola, WI. (Industry)
Organization: St Vincent's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB 77-04
Record Dates: First submitted 2005-07-19; First posted 2005-07-22 (Estimated); Last update posted 2006-06-27 (Estimated); Status verified 2005-07

CONDITIONS: Sleep Deprivation
Keywords: Diet; Chronic sleep deprivation; Weight; Cognitive impairment; Lipids; Inflammation; Resting metabolic rate; Weight Gain; Percent Body Fat; Hyperlipidemia
MeSH Terms: conditions — Sleep Deprivation; Body Weight; Cognitive Dysfunction; Inflammation; Weight Gain; Hyperlipidemias

INTERVENTIONS:
Drug: Controlled Dietary Intervention

SUMMARY:
The purpose of this study is to determine whether or not a low calorie, low glycemic index diet with omega-3 fatty acid supplements can prevent some of the negative consequences of sleep deprivation.

DETAILED DESCRIPTION:
This pilot study included 18 medical residents at two academic medical centers in New York City. All residents who participated in the study were assigned to work a night shift schedule for two weeks, and began the study on the morning prior to their first evening shift. The study subjects were randomly assigned to one of two groups:

* Intervention diet -- consisting of 40% carbohydrates, 30% protein, and 30% fat with 2.4g of long chain fatty acid supplements (n=9) Total calories for males was 1600/day, and 1200/day for females
* Control group -- ad lib diet.

Main outcome measures included:

* weight
* resting metabolic rate
* percent body fat
* lipid profile
* CRP
* fasting glucose and insulin levels
* urinary neurotransmitter levels
* salivary cortisol
* six cognitive tests of memory, attention, and executive function.

Subjects were tested on day 1, 7, and 14 of the study.

ELIGIBILITY:
Inclusion Criteria:

* Medical resident in good standing at Cabrini Medical Center or Saint Vincent's Hospital, NY.
* Must be scheduled for two consecutive weeks of night shift work.

Exclusion Criteria:

* Febrile illness
* Smoker
* Food allergies of any kind
* Taking any prescription medication
* History of diabetes or thyroid dysfunction
* Body mass index (BMI)>30
* Pregnancy

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18
Dates: Start 2004-09; Study Completion 2005-04

PRIMARY OUTCOMES:
Resting Metabolic Rate

SECONDARY OUTCOMES:
Weight
Percent Body Fat
Waist Circumference
Lipid Profile
C-reactive Protein Levels
Fasting serum glucose
Fasting serum insulin
Urinary neurotransmitter levels
Salivary a.m. cortisol levels
Cognitive scores on: Stroop Test, Hopkins Verbal Learning Test, Trail Making Test, Digit Span, Block Design, Dynamic Visual Acuity, Short Form 36

CONTACTS AND LOCATIONS:
Overall Officials: Valerie A Jones, MD, Principal Investigator — Saint Vincent's Hospital, Manhattan; Steven M Lascher, DVM, Study Director — Saint Vincent's Hospital, Manhattan
Locations (1):
- Saint Vincent's Hospital, New York, New York, United States

REFERENCES:
- See also: Saint Vincent's Hospital — http://www.svcmc.org